CLINICAL TRIAL: NCT06169488
Title: The Lumbar Interbody Fusion vs. Multidisciplinary Rehabilitation (LIFEHAB) Trial
Acronym: LIFEHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Haukeland University Hospital (Other); Vestre Viken Hospital Trust (Other); St. Olavs Hospital (Other); Unicare (Unknown)
Responsible Party: Principal Investigator, Kjersti Storheim, Senior researcher, professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 506009
Record Dates: First submitted 2023-11-22; First posted 2023-12-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain
Keywords: persisting; chronic; low back pain; MRI spectroscopy; multidisciplinary rehabilitation; lumbar fusion surgery; lumbar interbody fusion; TLIF; rehabilitation; ALIF; LIFEHAB
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not have access to information about participants' allocated treatment groups (lumbar interbody fusion or multidisciplinary rehabilitation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lumbar Interbody Fusion (LIF) (Experimental): Per center standard, the LIF procedure is done in one or two levels between the second lumbar vertebra and sacrum, as a transforaminal lumbar interbody fusion (TLIF) or anterior lumbar interbody fusion (ALIF). Stabilization with screws is mandatory. TLIF employs bilateral pedicle screws. ALIF uses either pedicle or intra-device screws.
  At least one surgeon must be proficient in both procedure and implants. TLIF requires visual aids (microscope/magnifying glasses) for precise disc preparation. In the TLIF procedure, surgeons will maximize bone implantation into the disc space, anteriorly, posteriorly, or both.
  If the disc space is too narrow for an interbody device, autologous bone grafting into the disc space (local, spongious, or both) with posterior pedicle screw fixation is accepted. Optional posterolateral autologous bone grafting is allowed, but no substitutes or osteoinductive proteins (e.g., BMP). Surgical drain is optional.
  Interventions: Procedure: Lumbar Interbody Fusion
- Multidisciplinary Rehabilitation (Active Comparator): Rehabilitation, guided by a team of experienced specialists in physical medicine and rehabilitation and physiotherapists trained in cognitive therapy, will direct the multidisciplinary treatment. Patients receive 2.5-5 hour sessions 2-4 days weekly over 3-5 weeks. Standardization is maintained through pre-study training for providers, including seminars, podcasts, videos, and lectures.
  Individual screenings start the process, leading to focused discussions on thoughts, feelings, behaviour, and physical symptoms. A plan for the rehabilitation process with clearly defined individual goals will be worked out and revised every week. The three components described within the framework of cognitive functional therapy will be a template for the implementation of the functional and physical rehabilitation, involving pain understanding, exposure with control, and lifestyle changes like physical activity, sleep, diet, stress management, and social engagement.
  Interventions: Behavioral: Multidisciplinary rehabilitation

INTERVENTIONS:
Procedure: Lumbar Interbody Fusion — Fusion of one or two lumbar levels with either a transforaminal lumbar interbody fusion (TLIF) or an anterior lumbar interbody fusion (ALIF) procedure.
  Arms: Lumbar Interbody Fusion (LIF)
Behavioral: Multidisciplinary rehabilitation — Outpatient multidisciplinary rehabilitation based on the treatment model described by Brox et al and Hellum et al consisting of a cognitive approach and supervised physical and functional training, but the protocol is somewhat compressed in terms of time and additionally updated in line with recent years' research in cognitive functional rehabilitation.
  Arms: Multidisciplinary Rehabilitation

SUMMARY:
The goal of this randomized controlled trial is to compare lumbar interbody fusion surgery with multidisciplinary rehabilitation in participants aged 20-65 years with persisting (≥ one year) low back pain. The main question it aims to answer is:

• Is lumbar fusion surgery superior to multidisciplinary rehabilitation in alleviating persisting low back pain?

Participants will be randomized to either lumbar interbody fusion surgery or a multidisciplinary rehabilitation program.

If randomized to lumbar fusion interbody surgery, the participants will:

* undergo radiologic examinations, including X-ray, MRI, and MRI spectroscopy
* provide blood samples at four intervals including postoperatively
* complete PROMs at five intervals
* have their activity monitored through the ActivePAL accelerometer
* undergo lumbar fusion surgery

If randomized to multidisciplinary rehabilitation, the participants will:

* undergo radiologic examinations, including X-ray, MRI, and MRI spectroscopy
* provide blood samples at three intervals
* complete PROMs at five intervals
* have their activity monitored through the ActivePAL accelerometer
* undergo multidisciplinary rehabilitation

DETAILED DESCRIPTION:
Background: Low back pain (LBP) is the number one cause of disability worldwide. Chronic LBP (cLBP), also referred to as persisting low back pain, is defined as low back pain lasting at least twelve weeks, with a lifetime prevalence of about 23%. It represents extensive individual, societal, and financial burdens.

The etiology of cLBP is multifactorial with complex pathogenesis, and only a small proportion of patients with disabling cLBP have a well-understood pathophysiological cause. Over the last several decades, the biopsychosocial model of LBP has been the standard approach. Accordingly, current clinical guidelines recommend treatments such as advice to stay active, exercise, reassurance and coping strategies, analgesic medications, and avoiding bed rest. The existing treatments, however, have only small to moderate effects, and 85-90% of patients do not receive a pathoanatomical diagnosis (National Institute for Health and Care Excellence (NICE)).

Many pathophysiological hypotheses for cLBP have been proposed (e.g., annular tear, disc herniation, loss of disc height, facet joint degeneration, and Modic changes). For example, it has been hypothesized that cLBP with Modic changes is caused by bacterial infection. A Danish trial reported that antibiotic treatment was superior to placebo in selected cLBP patients with focal vertebral bone marrow changes (Modic changes graded by MRI of the lumbar spine). However, the Norwegian AIM (Antibiotic In Modic changes) study did not support this finding. Nonetheless, intervertebral disc (IVD) degeneration is generally accepted as a relevant cause of cLBP, especially among surgeons treating the condition. An experimental study of cultured human nucleus pulposus cells showed that acidic pH caused an increase in several pro-inflammatory, neurotrophic, and pain-related factors. This upregulation of inflammatory substances may, in turn, induce the ingrowth of nerve fibers into degenerative IVDs, possibly explaining how discs can become painful. Therefore, one possible approach to diagnose painful IVDs could be to measure IVD pH levels by MRI spectroscopy (MRS). The local inflammation in degenerative IVD is correlated with a systemic inflammatory response that can be measured in serum samples and is related to symptoms. Recent developments in diagnostics and biomarkers in the field may improve patient selection and support an individually tailored treatment.

A few randomized controlled trials have compared lumbar spine fusion with non-operative treatment, finding similar improvements in pain and disability for both treatment alternatives. This has led to guidelines recommending non-operative treatment.

The researchers in the current project aim to improve treatment, develop refined diagnostic assessments, and explore potential biomarkers in a multicenter randomized controlled trial (RCT), adding level-one evidence to the subject.

The overall concept is to assess whether there is a difference in treatment effect between modern lumbar interbody fusion (LIF) and multidisciplinary rehabilitation (MRE) for patients with cLBP. The researchers aim to:

* Evaluate the effect of LIF versus MRE at one-year follow-up (FU).
* Evaluate the treatment effectiveness at two-year FU in the cohort of patients crossing over from one treatment arm to the other at one-year FU. (Primary and secondary outcome measures will be the same as those listed in sections 1 through 12 of the 'Outcome Measures' section.
* Evaluate the effect of LIF versus MRE at one-year FU on physical activity, sleep disturbances, and circadian rhythm.
* Evaluate whether baseline MRS biomarkers are associated with treatment response after LIF at one-year FU.
* Evaluate whether baseline MRS biomarkers are associated with treatment response after MRE at one-year FU.
* Evaluate whether MRS biomarkers are associated with molecular biomarkers in blood samples collected at three time points.
* Evaluate if molecular biomarkers can identify patients with improvement after LIF at one-year FU.
* Evaluate if molecular biomarkers can identify patients with improvement after MRE at one-year FU.
* Evaluate, if feasible, the correlation between MRS biomarkers and perioperative pH measurement of the IVD.
* Evaluate the cost-effectiveness of LIF versus MRE from baseline to one-year FU The spinal surgeons will screen participants for trial eligibility by predetermined inclusion- and exclusion criteria and ensure that necessary imaging examinations (MRI and X-ray) have been done per protocol.

Patients will be invited to trial participation if all the inclusion criteria and none of the exclusion criteria are satisfied. Patients who may be relevant study candidates are set up for a new appointment with another surgeon associated with the project so that each potential participant receives an individual assessment by two different surgeons, ensuring a thorough evaluation and sufficient reflection period for the patient. To avoid undue pressure to participate in the study, one of the treating surgeons who have assessed the patient at the outpatient clinic will provide information about the project, and obtaining informed consent will be done by an independent third party, for example, a study nurse, a representative from rehabilitation or another surgeon associated with the project. To ensure comprehensive and unbiased information regarding both trial arms, representatives from the MRE arm will also have a face-to-face or electronic meeting with potential trial participants before their inclusion. General consent, as well as specific consent to the neuroscientific biobank, will be obtained. However, consent to the neuroscience biobank is not mandatory for study participation. The participant will be issued copies of the letter informing about the trial and the signed informed consent(s).

Eligible patients will be allocated in a 1:1 ratio between LIF and MRE, using a computer randomization procedure stratified by center. Block size and allocation sequence generation details will be provided in a separate document unavailable to those who enroll patients or assign treatment. Following screening, eligible participants will be randomized in a continuous manner. Treatment initiation will occur within three months of randomization for both treatment groups.

Baseline data collection will include sociodemographic variables (age, gender, BMI, ethnicity, educational level, work status), as well as information on physical workload, leisure activities, smoking habits, emotional distress (assessed with Hopkins Symptom Checklist-25 [HSCL-25]), fear avoidance beliefs (FABQ), Örebro Musculoskeletal Pain Screening Questionnaire (Short-form), and cLBP history (including duration and prior treatments such as spinal surgery, physiotherapy, and chiropractic therapy). At baseline, we will ask all participants to report their smallest worthwhile reduction of pain and disability (in percent, not specified to measurement instrument), what treatment group they hope to be randomized to, and how well they expect to be at one-year FU (Likert scale (1-7)). We will further ask all investigators at baseline to report what treatment allocation they think would be best for the individual participant if they were not participating in a study and to rate (Likert scale (1-7)) how well they expect the participant to be at one-year FU given the randomization.

Baseline sick listing and subsequent sick listing at each FU consultation will include documentation of complete work absence and part-time absence.

Prospective participants must undergo radiological examinations before study inclusion, including MRI and plain radiographs for measuring pelvic spine parameters. The MRI and radiographs must be obtained within six months before the initiation of treatment.

Hematological parameters (leucocytes, thrombocytes, hemoglobin (Hb)), sedimentation rate, CRP, electrolytes (Na and K), and measures of kidney (creatinine) and liver function (ALAT) will be assessed and registered at baseline if allocated to LIF intervention. Functional comorbidity index will be reported at screening and serve as a screening tool for other relevant illnesses together with physical examination at baseline.

The study will be monitored by the Clinical Trial Unit at Oslo University Hospital according to the standard by NorCRIN and Good Clinical Practice. Adverse events and serious adverse events will be registered at all study FUs. The study will focus on monitoring specific adverse events in individuals allocated to the LIF intervention. These events include the following:

* Deep and superficial wound infection and rupture of the surgical wound
* Hardware mechanical complications with loosening of pedicle screws and interbody implants before bony fusion of the addressed lumbar level are evidenced.
* Improper hardware placement
* Wrong-level surgery
* Dural tears leading to spinal headaches and possibly a pseudo-meningocele
* Nerve root injury possibly leading to chronic neuropathic pain, palsy, and dysfunction of the muscles affected.
* Postoperative spinal hematoma necessitating an acute surgical evacuation
* Cauda equina compression that may lead to transient or permanent dysfunction of the urinary bladder and bowel function.
* Potentially life-threatening hemorrhage by iatrogenic injury to large pelvic vessels
* Iatrogenic injury to the ureter necessitating additional urologic procedures
* Bowel perforation in case of ALIF
* Retrograde ejaculation due to iatrogenic injury to the lumbar autonomous nervous system (ALIF) Monitoring for these adverse events will involve clinical examination, blood sample analysis (including parameters such as Hb, CRP, and leukocytes), and radiologic imaging such as CT scans and MRI.

Blood samples for DNA genotyping (Genomics), methylation (Epigenetics), and RNA sequencing (Transcriptomics) will be collected at baseline, 6- and 12-months FU from participants who have consented to participate in the genetic analysis component of the study. Participation is optional. Participants who do not wish to participate in the genetic research may still participate in the study.

The researchers will also, at baseline, 6- and 12 months, measure a panel of 40 cytokines by duplicate serum analysis with a 40-plex Pro Human Chemokine multi-bead assay. Samples that can be used to analyze suspected molecular biomarkers in the future will also be collected.

For all participants throughout the study, the investigator and study site personnel will collect data about healthcare resource utilization associated with medical encounters. The cost-benefit analysis of LIF versus MRE will be assessed by QUALYs derived from EQ-5D-5L and hospital and community treatment costs. The following data will be collected:

* LIF: Time in theatre, duration of surgery, blood loss and transfusions, number of surgeons, anesthesiologists, and nurses, implant costs, length of sick leave, use of non-operative treatment (i.e., physiotherapy, rehabilitation), additional visits to the GP, additional follow-ups including imaging outside the study protocol.
* MRE: Medical consultations at the general practitioner or other primary care treatment, additional diagnostic tests (e.g., X-ray, MRI, CT, laboratory tests), medications (e.g., pain relievers, muscle relaxants, anti-inflammatories, antidepressants), time spent at treatment facilities, staffing costs, travel expenses (for patients traveling to rehabilitation institution for every treatment day or session), accommodation costs (for patients staying at the rehabilitation institution during the treatment period) and sick leave.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female patients between 20 and 65 years of age with persistent low back pain of at least one year's duration at inclusion
2. Received non-operative treatment in line with national [50] and international [49] guidelines, including at least self-management, exercise, and physical therapy, without satisfactory effect before study enrolment
3. Back-related disability: ODI 30 - 60 points at baseline
4. Back pain > leg pain
5. One- or two-level disc degeneration between L2 and sacrum with any of the following:

   * High-intensity zone (HiZ)
   * Modic changes
   * Severe disc height reduction exceeding 50% of the cranial disc

Exclusion Criteria:

1. Multilevel disc degeneration requiring intervention beyond two levels
2. Spondylolysis or lytic spondylolisthesis
3. History of previous spondylodiscitis
4. Previous lumbar fusion surgery
5. Scoliosis >20 degrees
6. Signs of a vertebral fracture at the planned level of fusion or its adjacent levels
7. Active smokers
8. Unlikely to adhere to treatment or complete follow-up (e.g., ongoing serious psychiatric disease, drug abuse, plans to move outside the catchment areas of the trial centers)
9. Significant nerve root compression assessed by MRI and clinical examination
10. BMI > 40
11. Not understanding the Norwegian language.
12. Generalized myalgia, including history or signs of fibromyalgia and myalgic encephalitis
13. Contraindications to MRI (e.g., cardiac pacemaker electrodes, metal implants in the eye or brain, claustrophobia).
14. Active cancer
15. Disabling chronic neurological disease (e.g., Parkinson's disease, ALS, MS)
16. Disabling osteoarthritis of the hip or knee (Kellgren & Lawrence grade III or higher)
17. Daily use of morphine equivalents ≥ 60mg or regular use of morphine-containing pain patches
18. Decline specific treatment arm

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI): Change in percent | At one-year follow-up
  Improvement in the ODI score of a minimum of 30% from baseline. The ODI questionnaire examines the level of disability based on 10 everyday activities of daily living. Each item consists of 6 statements which are scored from 0 to 5, with 0 indicating the least disability and 5 the highest level of disability. The total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI): Dichotomized | At one-year follow-up
  ODI dichotomized as a Positive response: PASS (ODI≤22), i.e., participant reaches a Patient Acceptable Symptom State or a Negative response (ODI >22).
Oswestry Disability Index (ODI): Continuous | At one-year follow-up
  Change in ODI from baseline (continuous variable)
Numeric Rating Scale back pain (NRS back pain) | At one-year follow-up
  Change in NRS back pain from baseline (continuous variable). The NRS is a 11-point numeric scale ranging from '0' (e.g. "no pain") to '10' (e.g. "worst possible pain").
Numeric Rating Scale leg pain (NRS leg pain) | At one-year follow-up
  Change in NRS leg pain from baseline (continuous variable). The NRS is a 11-point numeric scale ranging from '0' (e.g. "no pain") to '10' (e.g. "worst possible pain").
Global perceived effect (GPE) | At one-year follow-up
  The GPE scale asks the participant to rate, on a 7 point Likert scale, how much their condition has improved or deteriorated. GPE 1-2 defined as success (completely recovered (1), much better (2)), GPE 3-5 defined as no change (somewhat better (3), no change (4), somewhat worse (5)), GPE 6-7 defined as worsening (much worse (6), worse than ever (7))
EuroQol-5 dimensions-5 levels (EQ-5D-5L) | At one-year follow-up
  Change in EQ-5D-5L from baseline (continuous variable). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each EQ-5D-5L dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Index scores range from -0.59 to 1, where1 is the best possible health state.
Fear Avoidance Beliefs Questionnaire (FABQ) | At one-year follow-up
  Change in FABQ from baseline (continuous variable). The questionnaire consists of 16 items in which a participant rates their agreement with each statement on a 7-point Likert scale, where 0 = completely disagree, 6 = completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Hopkins Symptom Check List (HSCL-25) | At one-year follow-up
  Change in HSCL-25 from baseline (continuous variable). The HSCL-25 consists of 25 items: Part I of the HSCL-25 has 10 items for anxiety symptoms; Part II has 15 items for depression symptoms. The scale for each question includes four categories of response ("Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively). Two scores are calculated: the total score is the average of all 25 items, while the depression score is the average of the 15 depression items.
Pain Catastrophizing Scale (PCS) | At one-year follow-up
  Change in PCS from baseline (continuous variable). The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Adverse Events of special interest (AESI) and Serious Adverse Events (SAEs) | During study period (two years)
  Incidence of AESI and SAEs
Occupational status and return to work | At one-year follow-up
  To evaluate the effect of LIF versus MRE on ability to work, the participants will be asked about their occupational status and return to work
ActivePAL accelerometer and sleep diary | At one-year follow-up
  To evaluate the effect of LIF versus MRE on physical activity, sleep disturbances, and circadian rhythm
MRI spectroscopy biomarkers: Change in ODI from baseline (continuous variable) | At one-year follow-up
  To evaluate whether baseline MRS biomarkers are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation measured by change in ODI from baseline (continuous variable). MRI spectroscopy biomarkers
  1: Trichotomized disc-specific NOCISCORE® for disc acidity (NOCI-, NOCImild, NOCI+).
  2. Total disc-specific NOCISCORE® (continuous 0-10)
  3. Normalized disc-specific NOCISCORE® (continuous 0-1)
  The trichotomized NOCISCORE® is based on the total vs the normalized NOCISCORES® and is calculated as previously published by standardized custom post-processing (NOCISCAN-LS®; Aclarion Inc.) of spectral feature disc data on acidic pain markers (alanine, lactic acid, propionic acid) in relation to structural integrity markers (carbohydrate/collagen and proteoglycan)
  Biomarker 1 will be used as the primary MRI spectroscopy biomarker for assessing the association between baseline disc acidity and treatment response.
MRI spectroscopy biomarkers: Change in NRS back pain from baseline (continuous variable) | At one-year follow-up
  To evaluate whether baseline MRS biomarkers are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation measured by change in NRS back pain from baseline (continuous variable). MRI spectroscopy biomarkers
  1: Trichotomized disc-specific NOCISCORE® for disc acidity (NOCI-, NOCImild, NOCI+).
  2. Total disc-specific NOCISCORE® (continuous 0-10)
  3. Normalized disc-specific NOCISCORE® (continuous 0-1)
  The trichotomized NOCISCORE® is based on the total vs the normalized NOCISCORES® and is calculated as previously published by standardized custom post-processing (NOCISCAN-LS®; Aclarion Inc.) of spectral feature disc data on acidic pain markers (alanine, lactic acid, propionic acid) in relation to structural integrity markers (carbohydrate/collagen and proteoglycan)
  Biomarker 1 will be used as the primary MRI spectroscopy biomarker for assessing the association between baseline disc acidity and treatment response.
MRI spectroscopy biomarkers: Change in NRS leg pain from baseline (continuous variable) | At one-year follow-up
  To evaluate whether baseline MRS biomarkers are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation measured by change in NRS leg pain from baseline (continuous variable). MRI spectroscopy biomarkers
  1: Trichotomized disc-specific NOCISCORE® for disc acidity (NOCI-, NOCImild, NOCI+).
  2. Total disc-specific NOCISCORE® (continuous 0-10)
  3. Normalized disc-specific NOCISCORE® (continuous 0-1)
  The trichotomized NOCISCORE® is based on the total vs the normalized NOCISCORES® and is calculated as previously published by standardized custom post-processing (NOCISCAN-LS®; Aclarion Inc.) of spectral feature disc data on acidic pain markers (alanine, lactic acid, propionic acid) in relation to structural integrity markers (carbohydrate/collagen and proteoglycan)
  Biomarker 1 will be used as the primary MRI spectroscopy biomarker for assessing the association between baseline disc acidity and treatment response.
MRI spectroscopy biomarkers: Improvement in the ODI score of a minimum 30% from baseline | At one-year follow-up
  To evaluate whether baseline MRS biomarkers are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation measured by improvement in the ODI score of a minimum 30% from baseline. MRI spectroscopy biomarkers
  1: Trichotomized disc-specific NOCISCORE® for disc acidity (NOCI-, NOCImild, NOCI+).
  2. Total disc-specific NOCISCORE® (continuous 0-10)
  3. Normalized disc-specific NOCISCORE® (continuous 0-1)
  The trichotomized NOCISCORE® is based on the total vs the normalized NOCISCORES® and is calculated as previously published by standardized custom post-processing (NOCISCAN-LS®; Aclarion Inc.) of spectral feature disc data on acidic pain markers (alanine, lactic acid, propionic acid) in relation to structural integrity markers (carbohydrate/collagen and proteoglycan)
  Biomarker 1 will be used as the primary MRI spectroscopy biomarker for assessing the association between baseline disc acidity and treatment response.
MRI spectroscopy biomarkers and molecular biomarkers | At baseline, 6-, and 12 months follow-up
  To evaluate the association between MRI spectroscopy and molecular biomarkers. See outcomes 14-17 for MRI spectroscopy description and outcomes 19-22 for cytokine description.
Molecular biomarkers: Change in ODI from baseline (continuous variable) | At one-year follow-up
  To evaluate whether serum inflammatory cytokines are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation on change in ODI from baseline (continuous variable). The unit of measure of cytokines is concentration.
Molecular biomarkers: Change in NRS back pain from baseline (continuous variable) | At one-year follow-up
  To evaluate whether serum inflammatory cytokines are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation on change in NRS back pain from baseline (continuous variable). The unit of measure of cytokines is concentration.
Molecular biomarkers: Change in NRS leg pain from baseline (continuous variable) | At one-year follow-up
  To evaluate whether serum inflammatory cytokines are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation on change in NRS leg pain from baseline (continuous variable). The unit of measure of cytokines is concentration.
Molecular biomarkers: Improvement in the ODI score of a minimum 30% from baseline | At one-year follow-up
  To evaluate whether serum inflammatory cytokines are associated with treatment response after lumbar interbody fusion or multidisciplinary rehabilitation on improvement in the ODI score of a minimum 30% from baseline. The unit of measure of cytokines is concentration.
Cost-effectiveness: EQ-5D-5L | At one-year follow-up
  To evaluate the cost-effectiveness of lumbar interbody fusion versus multidisciplinary rehabilitation on change in EQ-5D-5L from baseline (continuous variable).
Cost-effectiveness: Hospital costs | At one-year follow-up
  To evaluate the cost-effectiveness of lumbar interbody fusion versus multidisciplinary rehabilitation on hospital costs.
Cost-effectiveness: Community costs including sick leave | At one-year follow-up
  To evaluate the cost-effectiveness of lumbar interbody fusion versus multidisciplinary rehabilitation on community costs including sick leave
Cost-effectiveness: Co-interventions (pharmacological and non-pharmacological) | At one-year follow-up
  To evaluate the cost-effectiveness of lumbar interbody fusion versus multidisciplinary rehabilitation on co-interventions (pharmacological and non-pharmacological)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hellum, PhD, Principal Investigator — Oslo University Hospital, Division of Orthopedic Surgery, OUS Ullevål
Locations (5):
- Norway (5):
  - Vestre Viken Hospital, Drammen
  - Haukeland University Hospital, Hagavik
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Montgomery MW, Yawetz S, Levy BD, Loscalzo J. Back to the History. N Engl J Med. 2017 May 4;376(18):1783-1788. doi: 10.1056/NEJMcps1607608. No abstract available. PMID 28467866
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Bez M, Zhou Z, Sheyn D, Tawackoli W, Giaconi JC, Shapiro G, Ben David S, Gazit Z, Pelled G, Li D, Gazit D. Molecular pain markers correlate with pH-sensitive MRI signal in a pig model of disc degeneration. Sci Rep. 2018 Nov 26;8(1):17363. doi: 10.1038/s41598-018-34582-6. PMID 30478330
- [Background] Hancock MJ, Maher CG, Laslett M, Hay E, Koes B. Discussion paper: what happened to the 'bio' in the bio-psycho-social model of low back pain? Eur Spine J. 2011 Dec;20(12):2105-10. doi: 10.1007/s00586-011-1886-3. Epub 2011 Jun 25. PMID 21706216
- [Background] Albert HB, Kjaer P, Jensen TS, Sorensen JS, Bendix T, Manniche C. Modic changes, possible causes and relation to low back pain. Med Hypotheses. 2008;70(2):361-8. doi: 10.1016/j.mehy.2007.05.014. Epub 2007 Jul 10. PMID 17624684
- [Background] Albert HB, Sorensen JS, Christensen BS, Manniche C. Antibiotic treatment in patients with chronic low back pain and vertebral bone edema (Modic type 1 changes): a double-blind randomized clinical controlled trial of efficacy. Eur Spine J. 2013 Apr;22(4):697-707. doi: 10.1007/s00586-013-2675-y. Epub 2013 Feb 13. PMID 23404353
- [Background] Braten LCH, Rolfsen MP, Espeland A, Wigemyr M, Assmus J, Froholdt A, Haugen AJ, Marchand GH, Kristoffersen PM, Lutro O, Randen S, Wilhelmsen M, Winsvold BS, Kadar TI, Holmgard TE, Vigeland MD, Vetti N, Nygaard OP, Lie BA, Hellum C, Anke A, Grotle M, Schistad EI, Skouen JS, Grovle L, Brox JI, Zwart JA, Storheim K; AIM study group. Efficacy of antibiotic treatment in patients with chronic low back pain and Modic changes (the AIM study): double blind, randomised, placebo controlled, multicentre trial. BMJ. 2019 Oct 16;367:l5654. doi: 10.1136/bmj.l5654. PMID 31619437
- [Background] Gilbert HTJ, Hodson N, Baird P, Richardson SM, Hoyland JA. Acidic pH promotes intervertebral disc degeneration: Acid-sensing ion channel -3 as a potential therapeutic target. Sci Rep. 2016 Nov 17;6:37360. doi: 10.1038/srep37360. PMID 27853274
- [Background] Weber KT, Alipui DO, Sison CP, Bloom O, Quraishi S, Overby MC, Levine M, Chahine NO. Serum levels of the proinflammatory cytokine interleukin-6 vary based on diagnoses in individuals with lumbar intervertebral disc diseases. Arthritis Res Ther. 2016 Jan 7;18:3. doi: 10.1186/s13075-015-0887-8. PMID 26743937
- [Background] Deng X, Zhao F, Kang B, Zhang X. Elevated interleukin-6 expression levels are associated with intervertebral disc degeneration. Exp Ther Med. 2016 Apr;11(4):1425-1432. doi: 10.3892/etm.2016.3079. Epub 2016 Feb 16. PMID 27073460
- [Background] Hiyama A, Suyama K, Sakai D, Tanaka M, Watanabe M. Correlational analysis of chemokine and inflammatory cytokine expression in the intervertebral disc and blood in patients with lumbar disc disease. J Orthop Res. 2022 May;40(5):1213-1222. doi: 10.1002/jor.25136. Epub 2021 Jul 11. PMID 34191345
- [Background] Gornet MG, Peacock J, Claude J, Schranck FW, Copay AG, Eastlack RK, Benz R, Olshen A, Lotz JC. Magnetic resonance spectroscopy (MRS) can identify painful lumbar discs and may facilitate improved clinical outcomes of lumbar surgeries for discogenic pain. Eur Spine J. 2019 Apr;28(4):674-687. doi: 10.1007/s00586-018-05873-3. Epub 2019 Jan 4. PMID 30610465
- [Background] Brox JI, Nygaard OP, Holm I, Keller A, Ingebrigtsen T, Reikeras O. Four-year follow-up of surgical versus non-surgical therapy for chronic low back pain. Ann Rheum Dis. 2010 Sep;69(9):1643-8. doi: 10.1136/ard.2009.108902. Epub 2009 Jul 26. PMID 19635718
- [Background] Brox JI, Reikeras O, Nygaard O, Sorensen R, Indahl A, Holm I, Keller A, Ingebrigtsen T, Grundnes O, Lange JE, Friis A. Lumbar instrumented fusion compared with cognitive intervention and exercises in patients with chronic back pain after previous surgery for disc herniation: a prospective randomized controlled study. Pain. 2006 May;122(1-2):145-55. doi: 10.1016/j.pain.2006.01.027. Epub 2006 Mar 20. PMID 16545523
- [Background] Brox JI, Sorensen R, Friis A, Nygaard O, Indahl A, Keller A, Ingebrigtsen T, Eriksen HR, Holm I, Koller AK, Riise R, Reikeras O. Randomized clinical trial of lumbar instrumented fusion and cognitive intervention and exercises in patients with chronic low back pain and disc degeneration. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1913-21. doi: 10.1097/01.BRS.0000083234.62751.7A. PMID 12973134
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. 2001 Volvo Award Winner in Clinical Studies: Lumbar fusion versus nonsurgical treatment for chronic low back pain: a multicenter randomized controlled trial from the Swedish Lumbar Spine Study Group. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2521-32; discussion 2532-4. doi: 10.1097/00007632-200112010-00002. PMID 11725230
- [Background] Fairbank J, Frost H, Wilson-MacDonald J, Yu LM, Barker K, Collins R; Spine Stabilisation Trial Group. Randomised controlled trial to compare surgical stabilisation of the lumbar spine with an intensive rehabilitation programme for patients with chronic low back pain: the MRC spine stabilisation trial. BMJ. 2005 May 28;330(7502):1233. doi: 10.1136/bmj.38441.620417.8F. Epub 2005 May 23. PMID 15911537